CLINICAL TRIAL: NCT03586037
Title: An Open-label, Sequence-randomized, Three-period, Six-sequence, Multiple Dosing Crossover Clinical Trial to Evaluate the Pharmacokinetic Interaction Between AD-2011 and AD-2012 in Healthy Male Volunteers
Brief Title: Evaluating the Pharmacokinetic Interaction Between AD-2011 and AD-2012
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-201
Record Dates: First submitted 2018-05-28; First posted 2018-07-13 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Hyperlipidemias; Hypertension
MeSH Terms: conditions — Hyperlipidemias; Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Period 1: AD-2011 10/20mg QD Period 2: AD-2012 80mg QD Period 3: AD-2011 10/20mg + AD-2012 80mg QD
  Interventions: Drug: AD-2011 10/20 mg; Drug: AD-2012 80mg; Drug: AD-2011 10/20 mg + AD-2012 80mg
- Sequence 2 (Experimental): Period 1: AD-2011 10/20mg QD Period 2: AD-2011 10/20mg + AD-2012 80mg QD Period 3: AD-2012 80mg QD
  Interventions: Drug: AD-2011 10/20 mg; Drug: AD-2012 80mg; Drug: AD-2011 10/20 mg + AD-2012 80mg
- Sequence 3 (Experimental): Period 1: AD-2012 80mg QD Period 2: AD-2011 10/20mg + AD-2012 80mg QD Period 3: AD-2011 10/20mg QD
  Interventions: Drug: AD-2011 10/20 mg; Drug: AD-2012 80mg; Drug: AD-2011 10/20 mg + AD-2012 80mg
- Sequence 4 (Experimental): Period 1: AD-2012 80mg QD Period 2: AD-2011 10/20mg QD Period 3: AD-2011 10/20mg + AD-2012 80mg QD
  Interventions: Drug: AD-2011 10/20 mg; Drug: AD-2012 80mg; Drug: AD-2011 10/20 mg + AD-2012 80mg
- Sequence 5 (Experimental): Period 1: AD-2011 10/20mg + AD-2012 80mg QD Period 2: AD-2011 10/20mg QD Period 3: AD-2012 80mg QD
  Interventions: Drug: AD-2011 10/20 mg; Drug: AD-2012 80mg; Drug: AD-2011 10/20 mg + AD-2012 80mg
- Sequence 6 (Experimental): Period 1: AD-2011 10/20mg + AD-2012 80mg QD Period 2: AD-2012 80mg QD Period 3: AD-2011 10/20mg QD
  Interventions: Drug: AD-2011 10/20 mg; Drug: AD-2012 80mg; Drug: AD-2011 10/20 mg + AD-2012 80mg

INTERVENTIONS:
Drug: AD-2011 10/20 mg — AD-2011 10/20 mg tablet
Drug: AD-2012 80mg — AD-2012 80mg tablet
Drug: AD-2011 10/20 mg + AD-2012 80mg — AD-2011 10/20 mg + AD-2012 80mg tablet

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetic Interaction Between AD-2011 and AD-2012 in healthy male volunteers.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetic Interaction, safety and tolerability of the combination compared with the single administration of AD-2011 and AD-2012.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male between 19 and 50 years of age at the time of screening
* Weight between 50 kg and 90 kg and body mass index (BMI) between 18.0 kg/m2 and 27.0 kg/m2

Exclusion Criteria:

* Clinically significant disease or history of clinically significant disease such as liver, kidney, nervous system, respiratory, endocrine*hematologic, cardiovascular, urinary, psychiatric
* Gastrointestinal problem or history of gastrointestinal problem and history of gastrointestinal surgery
* AST, ALT values over than 1.5 times of ULN at screening
* HDL values less than 35 mg/dL
* A person who has a history of drug abuse or who has positive result for an abuse drug in a urine screening test

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration | pre-dose to 24 hours
  Cmax of the total ingredient of AD-2011 and AD-2012
Area under the plasma concentration versus time curve | pre-dose to 24 hours
  AUCtau of the total ingredient of AD-2011 and AD-2012

SECONDARY OUTCOMES:
Time to reach Cmax | pre-dose to 24 hours
  Tmax of the total ingredient of AD-2011 and AD-2012
Concentration | pre-dose to 24 hours
  Ctrough of the total ingredient of AD-2011 and AD-2012
Elimination half-life | pre-dose to 24 hours
  t1/2 of the total ingredient of AD-2011 and AD-2012
Clearance | pre-dose to 24 hours
  CL/F of the total ingredient of AD-2011 and AD-2012
Volume of distribution | pre-dose to 24 hours
  Vd/F of the total ingredient of AD-2011 and AD-2012
Number of participants with adverse events | From Day 1 up to Day 45
  Incidence rate of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huh KY, Lee SW, Lee SB, Kim KT, Jang IJ, Lee S. Pharmacokinetic Interaction Among Ezetimibe, Rosuvastatin, and Telmisartan. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1290-1296. doi: 10.1002/cpdd.926. Epub 2021 Mar 1. PMID 33647189